CLINICAL TRIAL: NCT03824366
Title: Pilot Study of Same-session MR-only Simulation and Treatment With MRI-guided Adaptive Palliative RadioTherapy (MAP-RT)
Brief Title: Same-session MR-only Simulation and Treatment With MRI-guided Adaptive Palliative RadioTherapy
Acronym: MAP-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201901172
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Malignancy; Metastasis; Hemoptysis; Gastrointestinal Bleeding; Pelvic Bleeding; Superior Vena Cava Syndrome; Mediastinal Disease
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Hemoptysis; Gastrointestinal Hemorrhage; Superior Vena Cava Syndrome; Mediastinal Diseases | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Volumetric MR imaging planning (Experimental): * All patients will undergo volumetric MR imaging on treatment days in positioning appropriate for the specific treatment site.
  * Patients will receive standard of care palliative radiation therapy
  Interventions: Device: Volumetric MR imaging; Radiation: Radiation therapy

INTERVENTIONS:
Device: Volumetric MR imaging — This will most frequently be supine with arms positioned so not in the way of treatment beams.
Radiation: Radiation therapy — -Standard of care

SUMMARY:
This proposed study is unique in that patients will not undergo computed tomography (CT) simulation at any point during their treatment course and will instead have same-session magnetic resonance (MR)-only simulation and treatment planning, on-table, using the adaptive radiotherapy (ART) workflow. In this manner, patients requiring urgent treatment could initiate treatment as early as the day of initial radiation oncology consultation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignancy (biopsy proven or high clinical suspicion with urgent/emergent clinical indications for palliative RT)
* Requires delivery of palliative radiation therapy for the treatment of painful metastasis, hemoptysis, gastrointestinal bleeding, pelvic bleeding, or superior vena cava syndrome/bulky mediastinal disease.
* At least 18 years of age.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Pregnant. Patients of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Medical contraindication to undergoing MR imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices). Participants who opted out of data sharing in the informed consent will not be included.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researches must provide a methodologically sound proposal. Proposals should be directed to kim.hyun@wustl.edu. To gain access, data requestors will need to sign a data access agreement and provide proof of appropriate regulatory approvals as necessary.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients would be considered evaluable for the study if they were able to be scheduled for radiation treatment per protocol.
Period: Overall Study
Arm/Group | Volumetric MR Imaging Planning
Started | 20
Completed | 16
Not Completed | 4
Not completed — Death | 1
Not completed — Previously unidentified metal artifact | 1
Not completed — Unable to tolerate lying flat on MR table | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Volumetric MR Imaging Planning
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 66 [28 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Same-session MRI-only Simulation as Defined as More Than 70% of Patients Receiving at Least 70% of Their Scheduled Treatment Fractions on the First On-table Attempt for Each Respective Fraction.
Time Frame: Completion of enrollment (approximately 29 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Volumetric MR Imaging Planning
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were tracked through 1 week following the last day of MRgRT, an average of 2 weeks.
Arm/Group | Volumetric MR Imaging Planning
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volumetric MR Imaging Planning (N=16)
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Death due to disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volumetric MR Imaging Planning (N=16)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03824366/Prot_SAP_000.pdf